CLINICAL TRIAL: NCT03292029
Title: Pilot Medical Evaluation of the T50 Calcification Inhibition Test in NephroCare Clinics
Brief Title: Pilot Medical Evaluation of the T50 Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HD-T50-01-ES
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Renal Failure; Cardiovascular Diseases; Vascular Calcification
Keywords: Renal replacement therapy; Haemodialsysis; Calcification Inhibition Test
MeSH Terms: conditions — Renal Insufficiency; Cardiovascular Diseases; Vascular Calcification

STUDY DESIGN:
Intervention Model Description: Exploratory, interventional, open, multi-center, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T50 Calcification Inhibition Test (CIT) (Other): Measurement of T50 CIT and fetuin-A serum values
  Interventions: Diagnostic Test: T50 Calcification Inhibition Test (CIT)

INTERVENTIONS:
Diagnostic Test: T50 Calcification Inhibition Test (CIT) — Measurement of predialysis T50 CIT and fetuin-A values in serum of hemodialysis patients

SUMMARY:
This pilot study aims to evaluate in an exploratory way the predictive power of a novel in vitro test (T50 Calcification Inhibition Test, T50 CIT), which measures the mineralization inhibition capacity of blood, in terms of its association with time to all-cause mortality in haemodialysis patients.

DETAILED DESCRIPTION:
Disturbances in mineral and bone metabolism centrally contribute to the exceedingly elevated risk for cardiovascular (CV) disease in dialysis patients. A novel in vitro test (T50 Calcification Inhibition Test, T50 CIT) has been developed, which measures the mineralization inhibition capacity of blood. This pilot study aims to exploratory examine the predictive power of baseline T50 CIT and fetuin-A (protein which is centrally involved in the inhibition of the formation of crystalline hydroxyapatite) values in terms of their association with all-cause mortality in an unselected cohort of haemodialysis patients. Moreover, the study shall investigate the association between baseline T50 CIT and fetuin-A values with CV related mortality, all-cause hospitalization and CV related hospitalization. Finally, the study aims to compare the predictive power of T50 CIT values with a set of six established calcification-related parameters (albumin, phosphate, calcium, magnesium, bicarbonate and fetuin-A). After baseline blood sampling the patients will be followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by study patient and investigator/authorised physician
* Minimum age of 18 years
* Incident and prevalent haemodialysis patients
* Three haemodialysis treatments per week

Exclusion Criteria:

* Any condition which could interfere with the patient's ability to comply with the study
* Pregnancy (pregnancy test will be conducted with female patients aged <= 55 years) or lactation period
* Participation in an interventional clinical study during the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
T50 CIT values | Baseline after signed informed consent
  The primary objective of this pilot study is to exploratory examine the predictive power of baseline T50 CIT values in terms of their association with time to all-cause mortality in haemodialysis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Rincon Bello, Dr., Principal Investigator — Fresenius Medical Care Spain
Locations (8):
- Spain (8):
  - Centro de Diálisis Barcelona - Glories, Barcelona
  - Centro de Diálisis Barcelona - Diagonal, Barcelona
  - Centro de Diálisis Barcelona - Rosselló, Barcelona
  - Centro de Diálisis Granollers, Granollers
  - Centro de Diálisis Hospitalet, L'Hospitalet de Llobregat
  - Centro de Diálisis Reus, Reus
  - Centro de Diálisis Tarragona, Tarragona
  - Centro de Diálisis Terrassa, Terrassa

REFERENCES:
- [Derived] Zawada AM, Wolf M, Rincon Bello A, Ramos-Sanchez R, Hurtado Munoz S, Ribera Tello L, Mora-Macia J, Fernandez-Robres MA, Soler-Garcia J, Aguilera Jover J, Moreso F, Stuard S, Stauss-Grabo M, Winter A, Canaud B. Assessment of a serum calcification propensity test for the prediction of all-cause mortality among hemodialysis patients. BMC Nephrol. 2023 Feb 15;24(1):35. doi: 10.1186/s12882-023-03069-6. PMID 36792998